CLINICAL TRIAL: NCT00765843
Title: A Randomized Controlled Trial of Custom Foot Orthoses for the Treatment of Plantar Heel Pain
Brief Title: A Trial of Custom Foot Orthoses for the Treatment of Plantar Heel Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rosalind Franklin University of Medicine and Science (Other)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Adam Fleischer, Assistant Professor, Rosalind Franklin University of Medicine and Science
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: ORT 067
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-06

CONDITIONS: Plantar Fasciitis
Keywords: heel pain
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Orthotic Devices; Foot Orthoses

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- custom foot orthoses (Active Comparator): Subjects will receive custom fabricated orthoses created from casts of the feet and according to individualized prescriptions. These orthoses are to be used in the standardized shoes provided to all subjects in the study.
  Interventions: Device: orthoses
- pre-fabricated orthoses (Active Comparator): Subjects will be provided pre-fabricated (non-customized) orthoses. These orthoses are to be used in the standardized shoes provided to all subjects in the study. for use in their shoes.
  Interventions: Device: orthoses
- sham insoles (Sham Comparator): Subjects will receive sham orthoses that are soft and pliable, but not designed to relieve pain. These orthoses are to be used in the standardized shoes provided to all subjects in the study.
  Interventions: Device: orthoses

INTERVENTIONS:
Device: orthoses — orthoses are provided for use in standardized shoes that all subjects receive
  Other Names: shoe insert

SUMMARY:
This is a study investigating treatment of plantar fasciitis (heel pain). Physicians commonly prescribe specialized orthoses (shoe inserts) to treat heel pain. This study will evaluate the reduction in heel pain associated with three types of orthoses. It is hypothesized that custom made orthoses will significantly decrease pain and improve foot function in comparison to prefabricated insoles and sham insoles.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included if they present for each of the following:

* Pain at plantar fascial attachment to calcaneal tubercle and/or pain distal from tubercle along plantar fascial band
* Typical post-static dyskinesia. Pain first steps in morning or when getting up after being seated for a period of time
* Patients will be ambulatory with an age range of 18-75 with plantar heel pain present for no more than one year.
* They will not have previous injection within 6 months or currently use prescription custom foot orthoses.
* Patient history, exam, x-rays, and ultrasound will rule out other etiologies of heel pain including proximal or local nerve entrapment, arthritis, bone cyst or tumor, or stress fracture. Since most patients will likely self-treat this condition prior to seeking care, the investigators will allow a washout period (appendix) and acetaminophen rescue analgesia provision.

Exclusion Criteria:

* Proximal musculoskeletal pathology (i.e., knee or hip arthritis, sciatica secondary to back pathology, significant limb length discrepancy.
* Use of gait assistive devices (crutches, canes, walkers).
* Inability to wear supportive closed toed shoes.
* Lack of range motion at the first metatarsophalangeal joint or subtalar joint.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2008-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Fleischer, DPM, MPH, Principal Investigator — Center for Lower Extremity Ambulatory Research (CLEAR)
Locations (2):
- United States (2):
  - Advocate Health Care, Chicago, Illinois
  - Scholl Foot and Ankle Center, North Chicago, Illinois

REFERENCES:
- See also: Center for Lower Extremity Ambulatory Research — http://www.CLEAR-Scholl.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Custom Foot Orthoses | Pre-fabricated Orthoses | Sham Insoles
Started | 26 | 25 | 26
Completed | 25 | 21 | 23
Not Completed | 1 | 4 | 3
Not completed — Lost to Follow-up | 1 | 3 | 2
Not completed — did not return to receive intervention | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Custom Foot Orthoses | Pre-fabricated Orthoses | Sham Insoles | Total
Number analyzed (Participants) | 26 | 25 | 26 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (13) | 51.3 (11) | 50.2 (12) | 49.6 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 16 | 49
  Male | 8 | 10 | 10 | 28
weight [Mean (Standard Deviation); unit: pounds] | 197.6 (42) | 187.4 (41) | 203.2 (49) | 196.2 (44)
height [Mean (Standard Deviation); unit: inches] | 65.8 (3.3) | 65.8 (3.4) | 66.2 (4.7) | 65.91 (3.8)
duration of plantar fasciitis [Mean (Standard Deviation); unit: months] | 4.9 (2.7) | 5.7 (3.6) | 5.7 (3.6) | 5.4 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Heel Pain
Description: Overall foot pain as determined by the Foot Function Index-Revised (FFI-R) survey. Foot pain is assessed by answering 11 questions regarding foot pain experienced over the past week. Scores may range from 11 to 66. Higher scores are indicative of greater foot pain.
Time Frame: baseline, one month and three months
Measure: Mean (Standard Deviation); unit: score on a survey
Arm/Group | Custom Foot Orthoses | Pre-fabricated Orthoses | Sham Insoles
Number analyzed (Participants) | 25 | 21 | 23
score on a survey
  baseline | 26.3 (8.6) | 27.9 (7.7) | 26.6 (9.3)
  one month | 23.9 (8.3) | 22.3 (6.5) | 19.1 (7.5)
  three months | 22.4 (9.0) | 23 (10.5) | 23.5 (8.9)
Statistical Analysis 1: Comparison: Custom Foot Orthoses vs Pre-fabricated Orthoses vs Sham Insoles; baseline comparisons; Test type: Superiority or Other; p = 0.78, ANOVA
Statistical Analysis 2: Comparison: Custom Foot Orthoses vs Pre-fabricated Orthoses vs Sham Insoles; one month comparisons; Test type: Superiority or Other; p = 0.21, ANOVA
Statistical Analysis 3: Comparison: Custom Foot Orthoses vs Pre-fabricated Orthoses vs Sham Insoles; three months comparisons; Test type: Superiority or Other; p = 0.93, ANOVA

ADVERSE EVENTS:
Arm/Group | Custom Foot Orthoses | Pre-fabricated Orthoses | Sham Insoles
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No